CLINICAL TRIAL: NCT04451629
Title: Effect of Exercise on Pain and Qulity of Life on People in Primary Dysmenorrhea Complaints
Brief Title: Effect of Exercise on Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SİNEM BAĞCI (Other)
Responsible Party: Sponsor-Investigator, SİNEM BAĞCI, Principal Investigator, Necmettin Erbakan University
Organization: Necmettin Erbakan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NEU
Record Dates: First submitted 2020-01-14; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Primary Dysmenorrhea
Keywords: Exercise; Quality of Life; Dysmenorrhea
MeSH Terms: conditions — Motor Activity; Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Parallel Assignment a experimental design with pre test and post test
Who Masked: Outcomes Assessor
Masking Description: Parallel Assignment a experimental design with pre test and post test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises group (Experimental): intervention group çalışma grubundaki kadın öğrencilere 8 hafta süresince haftada 4 kez 40 dakika boyunca pelvik taban ve core egzersizleri uygulatılacak
  Interventions: Behavioral: pelvıc base exercıse, core exercise
- control group (No Intervention): students will be watched without any intervention

INTERVENTIONS:
Behavioral: pelvıc base exercıse, core exercise — Effectıveness of the pelvıc base exercıse on the paın and qualıty of lıfe ın dysmenoral youth 40 minutes exercise intervention 4 times a week for 8 weeks
  Arms: Exercises group

SUMMARY:
Dismenored that menstruation is painful enough to interfere with the normal activity of the individual and require drug use. Dysmenorrhea is a localized pain in the lower abdominal quadrant and may spread to the back, waist, groin and vulva. This periodic pain may be accompanied by GIS complaints such as nausea, vomiting and frequent defecation, headache, emotional disorders and palpitations. Primary dysmenorrhea manifests itself as painful cramps in the lower part of the abdomen during the menstruation period without a pelvic pathology (endometriosis, pelvic adhesion or uterine fibroids, etc.). Menstrual problems affect 75% of adolescent girls and cause widespread medical treatment. The prevalence of primary dysmenorrhea in adolescents is significantly high, which is reported to be a major public health problem requiring attention. When Dysmenorrhea prevalence by examining the situation regarding in Turkey is noteworthy that dysmenorrhea prevalence in the 34-% 89.6% range. Non-drug applications are frequently used in the management of primary dysmenorrhea . Often, exercise is seen as an important method among these practices. Often, exercise is seen as an important method among these practices.

It has been reported that the effect of regular exercise on dysmenorrhea may be due to the effect of hormonal changes on the epithelial tissue of the uterus or an increase in endorphin levels, and it is concluded that dysmenorrhea reduces symptoms The aim of this study was to determine the effectiveness of pelvic floor exercise and quality of life in reducing pain in adolescents with primary dysmenorrhea.

DETAILED DESCRIPTION:
Research; planned as randomized controlled. The research is planned to be carried out in a faculty of Nursing, which provides service with 1 department of a university with 38.482 student capacity, continuing education with 15 faculties, 1,600 academic 1.152 administrative staff in the city center of Konya.

The population of the study is all female students who have been studying since 2018-2019 academic year. The population of the study is all female students who have been studying since 2018-2019 academic year.

The sample size of the study will be composed of female students who have the complaint of dysmenorrhea as a result of the pre-test and who agree to participate in the study.

The power analysis was used to determine the number of cases that required pelvic floor exercise and control groups for the study. In the study of Gamit et al., It was accepted that the mean pain decreased from 6.10 (1 ± 35) to 4.6 with a 1.5 decrease. Considering the data losses to be experienced during the study, 30 female patients were planned to be included in each group (Potur and Kömürcü 2014).

Working Group: Before randomization, Dismenorrhea Diagnosis Form will be applied to women students who agree to participate in the study according to the sample selection criteria and general information about the study will be given and their general consent will be obtained for participation in the study. In accordance with the sample size determined by power analysis, random assignment to experimental and control groups will be made. Block randomization system will be used.

Once randomization has occurred, it is not possible to blind the participants or health professionals. However, in the analysis phase of the data, the blind of the statistician and the writing of the report will be made.

Data Collection Technique and Tools Participation Criteria Form (Dysmenorrhea Diagnostic Form), Data Collection Form, Dysmenorrhea Follow-up Form, Visual Analogue Scale (VAS), Health Related Quality of Life Questionnaire (Short Form-36) (SF-36).

Data collection forms were created by the researcher in the light of literature .

ELIGIBILITY:
Inclusion Criteria:

* Describe dysmenorrhea pain severity as five and above on the visual comparison scale in the form of diagnosis of dysmenorrhea,

  * Being single,
  * Regular menstruation for the last 6 months (every 21-35 days with no intermittent bleeding),
  * Body Mass Index (BMI) is between 19-29,
  * 19-25 years of age
  * Voluntary acceptance of participation in the study

Exclusion Criteria:

* Having systemic and chronic diseases,
* Physical disability,
* Professional athlete,
* Using hormonal contraception (such as oral contraceptives and injections) and IUD,
* Secondary dysmenorrhea pathology (ultrasound examinations will be performed by a gynecologist).

Ages: 19 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Dysmenore as seen ın adolescent women face to face with the adolescent students themselves
Enrollment: 30 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2021-01-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (pain intensity) | 8 weeks
  Patients will be asked to keep a diary with VAS to determine the severity of pain during menstruation. Patients will be asked to mark their degree of pain on a horizontal line of 100 millimeters (mm). 0: no pain, 10: maximum means more pain than can be tolerated. The point marked on the line will be measured with a ruler and recorded as the pain intensity in cm during the menstruation. Patients will be asked to mark their pain on a separate scale for each day of menstruation. Cases will mark the most severe pain during the day during menstruation on the Visual Analogue Scale (VAS) during the 3 menstrual cycles in which the study is being conducted.8 weeks of application will be done and 3 cycle will be followed

SECONDARY OUTCOMES:
Quality of Life Questionnaire(short form-36)(SF-36) | 8 weeks
  SF-36 is a 36-item self-assessment scale consisting of eight subscales. This scale is based on physical function (10 items), role restrictions (physical (4 items) and emotional problems (3 items), pain (2 items), vitality (4 items), social function (2 items), mental health (5 items). and general health (5 items), each subscale is scored between 0-100 and 0 0 'is the lowest and "100' is the best quality of life.
  Before starting the study, the first measurement will be taken in the 2nd and 3rd menstrual cycle with an interval of 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Emel EGE, PROFESOR, Study Director — THESIS ADVISOR
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
will be planned with the conclusion of the study

REFERENCES:
- [Background] Abbaspour Z, Rostami M, Najjar S. Theeffect of exercise on primary dysmenorrhea. J Res Health Sci; 2006. 6(1):26-31.
- [Background] Apay SE, Arslan S, Akpinar RB, Celebioglu A. Effect of aromatherapy massage on dysmenorrhea in Turkish students. Pain Manag Nurs. 2012 Dec;13(4):236-40. doi: 10.1016/j.pmn.2010.04.002. Epub 2010 Sep 15. PMID 23158705
- [Background] Davis AR, Westhoff CL. Primary dysmenorrhea in adolescent girls and treatment with oral contraceptives. J Pediatr Adolesc Gynecol. 2001 Feb;14(1):3-8. doi: 10.1016/s1083-3188(00)00076-0. PMID 11358700
- [Background] Cakir M, Mungan I, Karakas T, Girisken I, Okten A. Menstrual pattern and common menstrual disorders among university students in Turkey. Pediatr Int. 2007 Dec;49(6):938-42. doi: 10.1111/j.1442-200X.2007.02489.x. PMID 18045301
- [Background] De Sanctis V, Soliman A, Bernasconi S, Bianchin L, Bona G, Bozzola M, Buzi F, De Sanctis C, Tonini G, Rigon F, Perissinotto E. Primary Dysmenorrhea in Adolescents: Prevalence, Impact and Recent Knowledge. Pediatr Endocrinol Rev. 2015 Dec;13(2):512-20. PMID 26841639
- [Background] Dixon JS, Bird HA. Reproducibility along a 10 cm vertical visual analogue scale. Ann Rheum Dis. 1981 Feb;40(1):87-9. doi: 10.1136/ard.40.1.87. PMID 7469530
- [Background] Erenel ŞA, Şentürk A. Sağlık Meslek Lisesi Öğrencilerinin Dismenore Yaşama Durumları ve Dismenore ile Baş Etmeye Yönelik Uygulamaları. Hacettepe Hemşirelik Yüksekokulu Dergisi. 2007. 2, 48-60.
- [Background] Erkek YZ, Pasinlioğlu T. Doğum Ağrısında Kullanılan Tamamlayıcı Tedavi Yöntemleri. Anadolu Hemşirelik ve Sağlık Bilimleri Dergisi, 2016. 19, 1.
- [Background] Gün Ç, Demirci N, Otrar M. Dismenore Yönetiminde Tamamlayıcı Alternatif Tedavileri Kullanma Durumu. Spatula DD, 2014. 4(4), 191-197.
- [Background] Doty E, Attaran M. Managing primary dysmenorrhea. J Pediatr Adolesc Gynecol. 2006 Oct;19(5):341-4. doi: 10.1016/j.jpag.2006.06.005. No abstract available. PMID 17060018
- [Background] Kapoor J, Kaur N, Sharma M, Kaur S. A study to assess the effectiveness of pelvic rocking exercises on dysmenorrhea among adolescent girls. International Journal of Applied Research. 2017. 3(3): 431-434.
- [Background] Khare D, Jain P. Effect of Different Exercise Techniques on Primary Dysmenorrhoea among Higher Secondary School Girls. International Journal of Science and Research (IJSR). Index Copernicus Value. 2015. 78-96.
- [Background] Mazza D. Primary dysmenorrhea. Women's Health Medicine. 2006. 3: 207-210.
- [Background] Potur DC, Komurcu N. The effects of local low-dose heat application on dysmenorrhea. J Pediatr Adolesc Gynecol. 2014 Aug;27(4):216-21. doi: 10.1016/j.jpag.2013.11.003. Epub 2014 Mar 19. PMID 24656704
- [Background] Rosyida DAC, Suwandono A, Ariyanti I, Suhartono, Mashoedi ID, Fatmasari D. Comparison of Effects of Abdominal Stretching Exercise and Cold CompressTherapy on Menstrual PainIntensity in Teenage Girls. Belitung Nursing Journal. 2017. 3(3):221-228.
- [Background] Sevil Ü. Adölesan Dönemi. İçinden: Kadın Sağlığı. Eds: Ahsen Şirin, Oya Kavlak. Bedray Basın Yayıncılık LtdŞti.,İstanbul.2008.s.57-91.
- [Background] Shahr-Jerdy S, Hosseini RS, Gh ME. The effect of stretching exercises on primary dysmenorrhea in adolescent girls. Biomedical Human Kinetics.2012; 4 : 127-132 .10.2478 / v10101-012-0024-y.
- [Background] Sutar A, Paldhikar S, Shikalgar N, Ghodey S. Effect of aerobic exercises on primary dysmenorrhoea in college students. IOSR Journal of Nursing and Health Science (IOSR -JNHS) ISSN: 2320-1959.p-Volume 5, Issue 5 Ver. V (Sep.Oct. 2016), PP 20-24.
- [Background] Taşkın L. (Ed). Doğum ve Kadın Sağlığı Hemşireliği. Üreme siklusus anomalileri. İçinde: X. baskı. Ankara: Sistem Ofset Matbaacılık; 2016:ss 733-736.
- [Result] Eryilmaz G, Ozdemir F, Pasinlioglu T. Dysmenorrhea prevalence among adolescents in eastern Turkey: its effects on school performance and relationships with family and friends. J Pediatr Adolesc Gynecol. 2010 Oct;23(5):267-72. doi: 10.1016/j.jpag.2010.02.009. Epub 2010 May 21. PMID 20493741
- [Result] Guvenc G, Kilic A, Akyuz A, Ustunsoz A. Premenstrual syndrome and attitudes toward menstruation in a sample of nursing students. J Psychosom Obstet Gynaecol. 2012 Sep;33(3):106-11. doi: 10.3109/0167482X.2012.685906. PMID 22901294
- [Result] Kannan P, Claydon LS. Some physiotherapy treatments may relieve menstrual pain in women with primary dysmenorrhea: a systematic review. J Physiother. 2014 Mar;60(1):13-21. doi: 10.1016/j.jphys.2013.12.003. Epub 2014 Apr 24. PMID 24856936
- [Result] Marsden JS, Strickland CD, Clements TL. Guaifenesin as a treatment for primary dysmenorrhea. J Am Board Fam Pract. 2004 Jul-Aug;17(4):240-6. doi: 10.3122/jabfm.17.4.240. PMID 15243011
- [Result] Nasir L, Bope ET. Management of pelvic pain from dysmenorrhea or endometriosis. J Am Board Fam Pract. 2004 Nov-Dec;17 Suppl:S43-7. doi: 10.3122/jabfm.17.suppl_1.s43. PMID 15575029
- [Result] Potur DC, Bilgin NC, Komurcu N. Prevalence of dysmenorrhea in university students in Turkey: effect on daily activities and evaluation of different pain management methods. Pain Manag Nurs. 2014 Dec;15(4):768-77. doi: 10.1016/j.pmn.2013.07.012. Epub 2013 Nov 11. PMID 24230963
- [Result] Seven M, Guvenc G, Akyuz A, Eski F. Evaluating dysmenorrhea in a sample of Turkish nursing students. Pain Manag Nurs. 2014 Sep;15(3):664-71. doi: 10.1016/j.pmn.2013.07.006. Epub 2014 Mar 14. PMID 24631318
- [Result] Motahari-Tabari N, Shirvani MA, Alipour A. Comparison of the Effect of Stretching Exercises and Mefenamic Acid on the Reduction of Pain and Menstruation Characteristics in Primary Dysmenorrhea: A Randomized Clinical Trial. Oman Med J. 2017 Jan;32(1):47-53. doi: 10.5001/omj.2017.09. PMID 28042403
- [Result] Ware JE Jr, Gandek B. Overview of the SF-36 Health Survey and the International Quality of Life Assessment (IQOLA) Project. J Clin Epidemiol. 1998 Nov;51(11):903-12. doi: 10.1016/s0895-4356(98)00081-x. PMID 9817107